CLINICAL TRIAL: NCT01644526
Title: A Pilot Study To Evaluate The CreatiVasc Hemoaccess Valve System In Patients Requiring Arteriovenous Graft Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An enhanced device has been developed
Sponsor: Diaxamed LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CVM-HVS-Phase I
Record Dates: First submitted 2012-04-03; First posted 2012-07-19 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: End Stage Renal Disease
Keywords: dialysis; vascular access; arteriovenous grafts; valve system
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hemoaccess Valve System (Experimental): Valve system for use with AV graft
  Interventions: Device: Hemoaccess Valve System

INTERVENTIONS:
Device: Hemoaccess Valve System — Device that allows blood to selectively flow into an arteriovenous graft to provide vascular access for dialysis then turn off the flow of blood to the graft in between dialysis sessions.

SUMMARY:
The ability to selectively control blood flow through an arteriovenous (AV) graft only when it is needed for dialysis may reduce the current repetitive complications such as thrombosis, venous hypertension post-dialysis bleeding, and blood steal from the extremities. The Hemoaccess Valve System (HVS) allows an AV graft to be turned on to blood flow when it is needed for dialysis then when dialysis is concluded, the device shuts off arterial blood flow and residual blood in the graft is flushed back into the body, using the dialysis blood lines. Once the graft is cleared of blood, the venous valve is then closed. Heparinized sterile saline reside in the graft between dialysis sessions. By having only saline in the graft and restoring normal blood flow to the artery and vein, it is believed that this will dramatically reduce the current complications associated with now having blood diverted through the graft 24/7.

DETAILED DESCRIPTION:
The Hemoaccess Valve System (HVS) is a subcutaneous valve device that is implanted when a new AV graft is placed. A saline pump delivers fluid to the arterial balloon valve and closes that end of the graft off to blood flow. Using the dialysis blood lines, saline flushes residual blood from the graft back into the body. Then the venous balloon valve closes and heparinized saline resides in the graft between dialysis sessions.

When the patient returns for dialysis, the dialysis technician deflates the valves and allows blood to flow to the graft for dialysis. (The saline inside the graft simply enters the blood stream.)

By only having saline inside the AV graft between dialysis sessions, there is no post-dialysis bleeding where the dialysis needles were cannulated, and because blood flow is restored to its normal course in the vein and artery, the traditional turbulent blood flow through the graft is eliminated, reducing the traditional complications caused when arterial blood is diverted through the graft then into the vein.

ELIGIBILITY:
Inclusion Criteria:

* Be a candidate for a new arteriovenous graft
* Be either currently on dialysis or ready to begin dialysis as soon as the access device (AV graft with Hemoaccess Valve System) is ready for use.
* Be prepared to receive dialysis at dialysis centers in proximity of study centers
* Have an outflow vein of greater than or equal to 3mm in diameter to which the graft can be successfully anastomosed.
* Be able to communicate with study personnel.
* Be considered by the physician to be readily available for subsequent visits.
* Be willing to comply with all aspects of the treatment and evaluation as directed over the duration of the study.
* Allow representatives of the Sponsor, the designated Clinical Research Organization, the Institutional Review Board and the FDA to review his/her relevant medical records that pertain to this study.

Exclusion Criteria:

* An identification of a central venous stenosis on the ipsilateral side is documented or otherwise identified
* An identification of an arterial venous stenosis on the ipsilateral side is documented or otherwise identified
* A hypercoagulable state is documented or otherwise identified and/or previous AV access failures have occurred without an identifiable cause.
* Has a life expectancy of less than one year.
* An immunodeficiency syndrome
* An organ transplant is expected within 6 months of enrollment
* 3 or more previous new AV graft or fistula placements have occurred.
* Body habitus (e.g., extremely small or obese arms( precludes HVS device implantation or access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Unassisted patency rate | 12 months
  Determine if the ability to limit blood flow to an AV graft only when it is needed for dialysis will increase unassisted patency rate of the test arm by a minimum of 50%. The New England Journal of Medicine study, "Effect of Dipyridamole plus Aspirin on Hemodialysis Graft Patency" (NEJM 360;21, 5/21/09) indicated a 1 year unassisted patency rate of 23% (77% required intervention). Our objective is to determine if the intervention rate can be reduced to 38-39% during the study, a 50% reduction in the expected intervention rate.

SECONDARY OUTCOMES:
Eliminate Post-Dialysis Needle Site Bleeding | 12 months
  Outcome measure: Reduce post-dialysis needle site bleeding by 95%.
  Currently most dialysis patients experience mild to severe post-dialysis bleeding when the large (15 gauge) dialysis needles are removed from their AV graft. The HVS device shuts off blood flow to the graft after dialysis therefore no post-dialysis bleeding should be experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Scribner, Study Director — CEO
Locations (1):
- Robert Scribner, Greenville, South Carolina, United States